CLINICAL TRIAL: NCT03365778
Title: An Educational Intervention to Increase Adoption of Selective Laser Trabeculoplasty as First-Line Treatment for Glaucoma
Brief Title: Educational Intervention to Adopt SLT as First-Line Glaucoma Treatment
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Wills Eye (Other)
Responsible Party: Principal Investigator, L. Jay Katz MD, Principal Investigator, Wills Eye
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: IRB # 17-641E
Record Dates: First submitted 2017-11-27; First posted 2017-12-07 (Actual); Results first posted 2020-01-30 (Actual); Last update posted 2020-01-30 (Actual); Status verified 2020-01

CONDITIONS: Primary Open-angle Glaucoma
Keywords: educational intervention; SLT; selective laser trabeculoplasty; POAG; eye drops; Primary Open Angle Glaucoma
MeSH Terms: conditions — Glaucoma, Open-Angle | interventions — Ophthalmologists

STUDY DESIGN:
Intervention Model Description: Selective Laser Trabeculoplasty (SLT) Educational Intervention group (n=20) or Usual Care group (n=20). Knowledge, beliefs, barriers, and attitudes about SLT vs. medication as first line treatment of glaucoma will be assessed in both groups.
  To evaluate barriers for widespread adoption of this procedure, we assessed beliefs and attitudes of ophthalmologists regarding SLT. We developed an educational slide presentation targeted at physicians to increase consideration of SLT earlier in glaucoma treatment paradigm.
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Patient Educational Intervention group (Active Comparator): Patients receive educational materials regarding selective laser trabeculoplasty (SLT) versus topical medication (ophthalmic eye drops) to lower eye pressure.
  Interventions: Other: Patient Educational Intervention
- Usual care group (Placebo Comparator): Patients receive standard of care.
  Interventions: Other: Usual Care
- Ophthalmologist Educational Intervention group (Other): General ophthalmologists, ophthalmology residents, and glaucoma specialists in the Wills Eye Hospital physician contact database receive online survey and educational slide presentation regarding selective laser trabeculoplasty (SLT).
  Interventions: Other: Ophthalmologist Educational Intervention

INTERVENTIONS:
Other: Patient Educational Intervention — Patients will respond to 5 questions regarding selective laser trabeculoplasty (SLT) versus topical medication to lower eye pressure. Then they will receive educational materials including 20 printed slides and view a 3 minute video on safety and efficacy of SLT. If patients agree to SLT, assistance in scheduling will be provided.
  Arms: Patient Educational Intervention group
Other: Usual Care — Patients will respond to 5 questions regarding selective laser trabeculoplasty (SLT) versus topical medication to lower eye pressure. No other guidance will be provided.
  Arms: Usual care group
Other: Ophthalmologist Educational Intervention — Responses to online survey regarding beliefs and attitudes towards selective laser trabeculoplasty (SLT) before and after educational slide presentation were recorded and compared between physician specialty groups.
  Other Names: Ophthalmologists
  Arms: Ophthalmologist Educational Intervention group

SUMMARY:
The purpose of this study is to develop an educational program that will help improve the patients' understanding of what laser treatment is, how it might be beneficial to them, and why it should be the first eye pressure lowering glaucoma treatment to consider before the use of glaucoma eye drops.

DETAILED DESCRIPTION:
Glaucoma is a disease characterized by optic nerve damage, visual field defects, elevated intraocular pressure (IOP) and progressive vision loss. More than 3 million Americans have glaucoma and more than 150,000 are blind as a result.

Regular use of glaucoma medications can usually lower intraocular pressure (IOP), prevent disease progression, preserve vision and prevent blindness. However, many people with glaucoma do not always use their medication as directed, with about one-third to one-half of patients with glaucoma not taking their drops as often as necessary, or have difficulty putting in the drops. There are also numerous local side effects from using glaucoma eye drops including red eyes, blurry vision and dry eye symptoms. Systemic side effects from eye drops range from triggering asthma, to lethargy and depression.

Selective laser trabeculoplasty (SLT) has been used safely and effectively for the treatment of elevated IOP in patients with open angle glaucoma for more than 20 years. SLT may result in mild and temporary IOP elevation, but this is a small risk and rarely significant. Other side effects include blurred vison and inflammation of the cornea (front, clear part of the eye), but they are extremely rare.

The purpose of this study is to develop an educational program that will help improve the patients' understanding of what laser treatment is, how it might be beneficial to them, and why it should be considered as first glaucoma treatment before the use of glaucoma eye drops.

ELIGIBILITY:
Inclusion Criteria:

* patients between 40 and 90 years of age
* high-risk ocular hypertension, primary open-angle glaucoma, or pseudo-exfoliation glaucoma
* currently treated with at least one glaucoma eye drop with stable intraocular pressure

Exclusion Criteria:

* previous laser trabeculoplasty
* previous glaucoma surgery

Ages: 40 Years to 90 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2017-10-23 (Actual); Primary Completion 2018-12-01 (Actual); Study Completion 2019-12-31 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: L. Jay Katz, MD, Principal Investigator — Wills Eye
Locations (1):
- Wills Eye Hospital, Philadelphia, Pennsylvania, United States

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Tran E, Sanvicente C, Hark LA, Myers JS, Zhang Q, Shiuey EJ, Tran J, Bonafede L, Hamershock RA, Withers C, Katz LJ. Educational intervention to adopt selective laser trabeculoplasty as first-line glaucoma treatment: Randomized controlled trial: Educational intervention on selective laser trabeculoplasty. Eur J Ophthalmol. 2022 May;32(3):1538-1546. doi: 10.1177/11206721211018365. Epub 2021 May 27. PMID 34041935

RESULTS

PARTICIPANT FLOW:
Groups:
- Patient Educational Intervention Group: Patients receive educational materials regarding selective laser trabeculoplasty (SLT) versus topical medication (ophthalmic eye drops) to lower eye pressure.
  Educational intervention: Patients will respond to 5 questions regarding selective laser trabeculoplasty (SLT) versus topical medication to lower eye pressure. Then they will receive educational materials including 20 printed slides and view a 3 minute video on safety and efficacy of SLT. If patients agree to SLT, assistance in scheduling will be provided.
- Ophthalmologist Educational Intervention Group: General ophthalmologists, ophthalmology residents, and glaucoma specialists in the Wills Eye Hospital physician contact database received an online survey and educational slide presentation regarding selective laser trabeculoplasty (SLT).
Period: Overall Study
Arm/Group | Patient Educational Intervention Group | Usual Care Group | Ophthalmologist Educational Intervention Group
Started | 16 | 17 | 53
Completed | 16 | 17 | 53
Not Completed | 0 | 0 | 0

BASELINE CHARACTERISTICS:
Population: Ophthalmologists were sent selective laser trabeculoplasty (SLT) educational information and online survey access only. They did not provide personal information such as date of birth, gender, ethnicity, race. Baseline characteristics in this group only include number of general ophthalmologists, ophthalmology residents and glaucoma specialists.
Groups:
- Ophthalmologist Educational Intervention Group: General ophthalmologists, ophthalmology residents, and glaucoma specialists in the Wills Eye Hospital physician contact database received online survey and educational slide presentation regarding selective laser trabeculoplasty (SLT). No other personal information i.e. age, gender, ethnicity, race was provided by these participants.
- Total: Total of all reporting groups
Arm/Group | Patient Educational Intervention Group | Usual Care Group | Ophthalmologist Educational Intervention Group | Total
Number analyzed (Participants) | 16 | 17 | 53 | 86
Age, Categorical [Count of Participants; unit: Participants] — Population: Ophthalmologists did not provide personal information such as date of birth, gender, ethnicity, race. Baseline characteristics in this group only include number of general ophthalmologists, ophthalmology residents and glaucoma specialists.
  Participants
    number analyzed (Participants) | 16 | 17 | 0 | 33
    <=18 years | 0 | 0 |  | 0
    Between 18 and 65 years | 8 | 8 |  | 16
    >=65 years | 8 | 9 |  | 17
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Ophthalmologists did not provide personal information such as date of birth, gender, ethnicity, race. Baseline characteristics in this group only include number of general ophthalmologists, ophthalmology residents and glaucoma specialists.
  Participants
    number analyzed (Participants) | 16 | 17 | 0 | 33
    Female | 8 | 7 |  | 15
    Male | 8 | 10 |  | 18
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 1 | 1 | 0 | 2
  Not Hispanic or Latino | 9 | 14 | 0 | 23
  Unknown or Not Reported | 6 | 2 | 53 | 61
Race (NIH/OMB) [Count of Participants; unit: Participants]
  American Indian or Alaska Native | 0 | 0 | 0 | 0
  Asian | 1 | 0 | 0 | 1
  Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0
  Black or African American | 5 | 13 | 0 | 18
  White | 5 | 2 | 0 | 7
  More than one race | 0 | 0 | 0 | 0
  Unknown or Not Reported | 5 | 2 | 53 | 60
Region of Enrollment [Number; unit: participants]
  United States | 16 | 17 | 53 | 86
Type of Ophthalmologist [Count of Participants; unit: Participants] — Ophthalmologists participated in SLT educational presentation and online survey. Baseline characteristics collected from this group only include type of ophthalmologist. Age, gender, ethnicity and race were not captured. Population: Patient Educational Intervention and Usual Care Groups are not compared in Type of Ophthalmologist baseline data.
  Participants
    General ophthalmologists: number analyzed (Participants) | 0 | 0 | 53 | 53
    General ophthalmologists | 0 | 0 | 26 | 26
    Ophthalmology Residents: number analyzed (Participants) | 0 | 0 | 53 | 53
    Ophthalmology Residents | 0 | 0 | 5 | 5
    Glaucoma Specialists: number analyzed (Participants) | 0 | 0 | 53 | 53
    Glaucoma Specialists | 0 | 0 | 22 | 22

OUTCOME MEASURES:

1. Primary Outcome: Completion of Selective Laser Trabeculoplasty (SLT)
Description: Percentage of patients who elect the Selective Laser Trabeculoplasty (SLT), as treatment for lowering eye pressure, compared between a group receiving SLT Educational Intervention and a Usual Care group. Follow-up eye examinations will be screened for a 6-month period to assess number of completed SLTs.
Time Frame: 1 hour
Measure: Count of Participants; unit: Participants
Groups:
- Educational Intervention Group: Patients receive educational materials regarding selective laser trabeculoplasty (SLT) versus topical medication (ophthalmic eye drops) to lower eye pressure.
  Educational intervention: Patients will respond to 5 questions regarding selective laser trabeculoplasty (SLT) versus topical medication to lower eye pressure. Then they will receive educational materials including 20 printed slides and view a 3 minute video on safety and efficacy of SLT. If patients agree to SLT, assistance in scheduling will be provided.
Arm/Group | Educational Intervention Group | Usual Care Group
Number analyzed (Participants) | 16 | 17
Participants | 10 | 6

2. Primary Outcome: Measure Educational Effects of Selective Laser Trabeculoplasty (SLT)
Description: Attitudes were assessed in the Patient Educational Intervention group before and immediately following intervention to determine how receptive they were regarding Selective Laser Trabeculoplasty (SLT) as a therapy to lowering eye pressure as compared to the more common therapy of daily eye drops.
Time Frame: 1 hour
Population: Usual Care group not included since they did not receive education intervention.
Measure: Count of Participants; unit: Participants
Arm/Group | Educational Intervention Group | Usual Care Group
Number analyzed (Participants) | 16 | 0
Participants
  Pre-Intervention Yes | 0 | 0
  Post-Intervention Yes | 12 | 0

3. Secondary Outcome: Measure Educational Effects of Selective Laser Trabeculoplasty (SLT) Among Ophthalmologists
Description: To evaluate barriers for widespread adoption of selective laser trabeculoplasty (SLT) as first line treatment of high eye pressure, we assessed the beliefs and attitudes of ophthalmologists regarding SLT. An educational slide presentation and survey targeted physicians to increase awareness and consideration of SLT earlier in the glaucoma treatment paradigm. Number of respondents who currently offer laser treatment for newly diagnosed glaucoma patients.
Time Frame: 30 minutes
Measure: Count of Participants; unit: Participants
Arm/Group | Ophthalmologist Educational Intervention Group
Number analyzed (Participants) | 53
Participants | 45

ADVERSE EVENTS:
Time Frame: 1 hour
Groups:
- Usual Care Group: Patients receive standard of care and will respond to 5 questions regarding selective laser trabeculoplasty (SLT) versus topical medication to lower eye pressure. No other guidance will be provided.
Arm/Group | Patient Educational Intervention Group | Usual Care Group | Ophthalmologist Educational Intervention Group
All-Cause Mortality (participants affected / at risk) | 0/16 | 0/17 | 0/53
Serious Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/53
Other Adverse Events (participants affected / at risk) | 0/16 | 0/17 | 0/53

LIMITATIONS AND CAVEATS:
Questionnaires limited determining how much attitudes changed immediately following education.

Small sample size limited ability to show significant differences. Location created difficulty in finding patients that fit inclusion criteria.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (3):
  • Study Protocol and Statistical Analysis Plan (2017-06-01): https://cdn.clinicaltrials.gov/large-docs/78/NCT03365778/Prot_SAP_000.pdf
  • Informed Consent Form: Informed Consent Form for Patients (2017-06-15): https://cdn.clinicaltrials.gov/large-docs/78/NCT03365778/ICF_001.pdf
  • Informed Consent Form: Informed Consent Form for Ophthalmologists (2017-07-11): https://cdn.clinicaltrials.gov/large-docs/78/NCT03365778/ICF_002.pdf